CLINICAL TRIAL: NCT02172898
Title: Alcoholic Hepatitis: A Multicenter, Observational Study by the TREAT Consortium
Status: Completed | Type: Observational
Sponsor: Indiana University (Other)
Collaborators: National Institute on Alcohol Abuse and Alcoholism (NIAAA) (NIH)
Responsible Party: Principal Investigator, Naga P. Chalasani, Naga Chalasani, MD, FACG, Indiana University
Other Study IDs: TREAT Observational; U01AA021840-01 (NIH)
Record Dates: First submitted 2014-06-09; First posted 2014-06-24 (Estimated); Last update posted 2020-02-11 (Actual); Status verified 2020-02

CONDITIONS: Alcoholic Hepatitis
MeSH Terms: conditions — Hepatitis, Alcoholic

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — serum/plasma, peripheral mononuclear cells, genomic DNA, stool samples, urine, and liver tissue (where available)
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- Heavily Drinking Controls: Heavy alcohol drinking will be defined as > 40 grams per day on average in women and > 60 grams per day on average in men for a minimum of 6 months and within the 6 weeks prior to study enrollment. Heavy drinkers, who have just become abstinent within prior 2 weeks, including those we convince to seek treatment as part of the recruiting process, are eligible for enrollment. Control subjects must meet the following criteria: (1) AST, ALT, and total bilirubin levels must be within normal range; (2) no prior history of known alcoholic liver disease; and (3) absence of hepatosplenomegaly (from physical examination or radiographic imaging) or stigmata of liver disease.
- Subjects with AH: Diagnosis of AH will be established on published criteria based on history of heavy alcohol consumption (defined as > 40 grams per day on average in women and > 60 grams per day on average for men for a minimum of 6 months and within the 6 weeks prior to study enrollment), clinical evaluation and appropriate laboratory testing (as defined as total bilirubin > 2 mg/dL and AST > 50 U/L). When diagnosis of AH remains in question, a liver biopsy (if clinically feasible and subject has no contraindications) will be required. We plan to enroll patients with AH in special population infected with hepatitis B (HBV), hepatitis C (HCV), or HIV.

SUMMARY:
To conduct a prospective, multicenter, observational study of patients with well-characterized alcoholic hepatitis (AH) and frequency matched individuals (by age, gender, and race) with comparable history of alcohol consumption but no clinical evidence of liver disease (controls). At the end of the study, a robust clinical information, central bio-repository will be developed from both cases and controls.

ELIGIBILITY:
CASES: Heavy drinkers with alcoholic hepatitis

Inclusion criteria

1. The diagnosis of AH will be established on published criteria this is based on:

1. Average daily ethanol consumption of > 40 grams/day for women and > 60 grams/day for men for a minimum of 6 months and within the 6 weeks prior to study enrolment. Judgment regarding daily and yearly alcohol use will be made by the site investigator
2. Clinical evaluation and appropriate laboratory testing as defined by total bilirubin > 2 mg/dL and AST > 50 U/L. When the diagnosis of AH remains in question, a liver biopsy (if clinically feasible and that subject has no contra-indications) will be required.
3. Subjects with HBV, HCV and/or HIV will be eligible for enrollment

Exclusion criteria

1. Evidence of other liver diseases such as autoimmune or drug-induced
2. Significant concomitant medical illnesses such as uncontrolled congestive heart failure or COPD, or multiorgan failure
3. Abstinence of alcohol use > 6 weeks immediately preceding enrollment
4. Hemochromatosis
5. Wilson Disease
6. Active intravenous drug use

CONTROLS: Heavy drinkers without alcoholic hepatitis

Inclusion criteria

1. Average daily ethanol consumption of > 40 grams /day for women and > 60 grams/day for males for a minimum of 6 months and within the 6 weeks prior to study enrollment. In addition, heavy drinkers who have just become abstinent within prior 2 weeks are eligible to be enrolled. Judgment regarding daily and yearly alcohol use will be made by the site investigator
2. AST and ALT ≤ 50 and total bilirubin levels within normal range. If bilirubin is increased due to a suspected Gilbert's Syndrome, patient may be enrolled if the direct bilirubin is within normal limits

Exclusion criteria

1. Evidence of liver disease
2. Significant concomitant medical illnesses such as uncontrolled congestive heart failure or COPD, or multiorgan failure
3. Abstinence of alcohol use > 2 weeks immediately preceding enrollment
4. Hemochromatosis
5. Wilson Disease
6. Active intravenous drug use
7. Prior history of known alcoholic liver disease
8. Presence of hepatosplenomegaly from the physical examination/radiographic imaging or stigmata of liver disease

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Individuals with AH and suitable controls will be enrolled at Indiana University and affiliated hospitals. In addition, the enrollment will be conducted simultaneously at Mayo Clinic and Virginia Commonwealth University with the same target enrollment.
Sampling Method: Non-Probability Sample
Enrollment: 454 (Actual)
Dates: Start 2013-06 (Actual); Primary Completion 2018-06-29 (Actual); Study Completion 2019-07 (Actual)

PRIMARY OUTCOMES:
Developing a repository of biological samples from AH patients and heavy drinking controls. | Up to 1 year
  To conduct a prospective, multicenter, observational study of patients with well-characterized AH and frequency matched individuals (by age, gender, and race) with comparable history of alcohol consumption but no clinical evidence of liver disease (controls). At the end of the study, a robust clinical information, central bio-repository of serum/plasma, peripheral mononuclear cells, genomic DNA, stool samples, urine, and liver tissue (where available) will be developed from both cases and controls.

SECONDARY OUTCOMES:
Characterizing AH subjects and controls to serve as the foundation for novel mechanistic and therapeutic studies. | Up to 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Naga Chalasani, MD, Principal Investigator — Indiana University
Locations (2):
- United States (2):
  - Mayo Clinic, Rochester, Minnesota
  - Virginia Commonwealth University, Richmond, Virginia

REFERENCES:
- [Derived] Madathanapalli A, Tang Q, Lammert C, Samala N, Shah VH, Sanyal A, Chalasani N, Desai AP. Health-related quality of life is dynamic in alcoholic hepatitis and responds to improvement in liver disease and reduced alcohol consumption. Alcohol Clin Exp Res. 2022 Feb;46(2):252-261. doi: 10.1111/acer.14756. Epub 2021 Dec 16. PMID 34862610
- [Derived] Mathur K, Vilar-Gomez E, Connelly MA, He H, Sanyal AJ, Chalasani N, Jiang ZG. Circulating high density lipoprotein distinguishes alcoholic hepatitis from heavy drinkers and predicts 90-day outcome: lipoproteins in alcoholic hepatitis. J Clin Lipidol. 2021 Nov-Dec;15(6):805-813. doi: 10.1016/j.jacl.2021.10.002. Epub 2021 Oct 20. PMID 34756674
- [Derived] Shamseddeen H, Madathanapalli A, Are VS, Shah VH, Sanyal AJ, Tang Q, Liang T, Gelow K, Zimmers TA, Chalasani N, Desai AP. Changes in Serum Myostatin Levels in Alcoholic Hepatitis Correlate with Improvement in MELD. Dig Dis Sci. 2021 Sep;66(9):3062-3073. doi: 10.1007/s10620-020-06632-5. Epub 2020 Oct 19. PMID 33074470